CLINICAL TRIAL: NCT04250922
Title: A Randomized, Double-blind, Placebo-controlled Adjuvant Trial in Newly Diagnosed Primary Glioblastoma Subjects to Assess the Efficacy and Safety of LAM561 in Combination With Radiotherapy and Temozolomide Standard of Care Treatment.
Brief Title: LAM561 With RT and TMZ for Adults With Glioblastoma
Acronym: CLINGLIO
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laminar Pharmaceuticals (Industry)
Collaborators: Laboratory Corporation of America (Industry); Northern Institute for Cancer Research, Newcastle (Unknown); Theradis pharma (Unknown); LIPODOM THERAPEUTICS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIN-003-1806
Record Dates: First submitted 2019-06-18; First posted 2020-01-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Primary Glioblastoma; Glioblastoma Multiforme
Keywords: malignant
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, 2 parallel arms (1:1), adjuvant trial to assess the efficacy of LAM561 vs placebo in patients with ndGBM. The 2 arms are: Arm A: SoC + placebo for LAM561; Arm B: SoC + 12g/day of LAM561
  Treatment consists of 3 phases:
  1. Chemoradiotherapy (6 to 7 weeks)
     * RT in daily fractions of 2Gy, 5 days per week (60Gy)
     * TMZ 75mg/m2 daily (maximum of 49 days)
     * Placebo or LAM561 for 4 weeks (from week 3 to week 6, both inclusive) -Washout period (4 weeks)
  2. Maintenance (4-week cycles, maximum of 6 cycles)
     * Placebo/LAM561 daily in the first 3 weeks of each cycle, followed by 7 days washout
     * TMZ 150-200mg/m2 daily in the first 5 days of each cycle
  3. Monotherapy: 4-week cycles until disease progression, unacceptable toxicity or lack of clinical benefit Placebo/LAM561 daily in the first 3 weeks of each cycle followed by 7 days washout
Who Masked: Participant, Care Provider, Investigator
Masking Description: At the Screening Visit, the IRT will assign a unique number to the subject. The site will use the IRT to receive drug kit numbers and a unique randomization number.
  Subjects will be randomized to Arm A or B in a 1:1 ratio. Drug kit numbers and treatment content will be assigned according to a list generated before the start of the study. At interim, the IRT vendor will transfer the list of attribution to the iSCs. After the final lock, the list of attribution will be transmitted to the company involved in analysis. The IRT vendor will be in charge of the stock management/logistics in each site and shipments. Upon receipt of study drug, the study site will acknowledge receipt in the IRT system.
  The investigators, the study site personnel and subject will remain blinded to throughout the course of the study. The IRT will provide access to for a subject in case of medical emergency. If sponsor/clinical team should break the blind, the reason will be documented on the eCRF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: SoC + placebo for LAM561 (Placebo Comparator): Chemoradiation Phase: all subjects undergo focal RT, with a treatment given 5 days per week over ~6 weeks (no more than 7 weeks). TMZ will be administered at 75 mg/m2 orally, once daily, continuously throughout the RT for a maximum of 49 days. Subjects in Arm A will receive placebo every day from Day 1 of week 3 to the end of this Phase.
  The start of the first cycle during the Maintenance (Adjuvant) Phase will be scheduled ~28 days (and never more than 42 days) after the last day of chemoradiation. During the Maintenance Phase, subjects will receive oral TMZ 150-200 mg/m2 once daily on Days 1-5 of each 28-day cycle for 6 cycles.
  Subjects in Arm A will receive placebo every day during the first 3 weeks of each 28-day cycle and until progression. Patients will continue with Placebo after cycle 6 of the monotherapy phase until end of study. Adjuvant treatment will be discontinued upon determination of tumour progression, unacceptable toxicity or refusal to continue study treatment.
  Interventions: Drug: TMZ; Radiation: RT
- Arm B: SoC + 12 g/day of LAM561 (Experimental): Chemoradiation Phase: all subjects undergo focal RT, with a treatment given 5 days per week over ~6 weeks (no more than 7 weeks). TMZ will be administered at 75 mg/m2 orally, once daily, continuously throughout the RT for a maximum of 49 days. Subjects in Arm B will receive LAM561 every day from Day 1 of week 3 to the end of this Phase.
  The start of the first cycle during the Maintenance Phase will be scheduled ~28 days (and never more than 42 days) after the last day of chemoradiation. During the Maintenance Phase, subjects will receive oral TMZ 150-200 mg/m2 once daily on Days 1-5 of each 28-day cycle for 6 cycles.
  Subjects in Arm B will receive LAM561 during the Maintenance Phase. Patients will continue to be administered with LAM561 after cycle 6 of the monotherapy phase until end of study. Adjuvant treatment will be discontinued upon determination of tumour progression, unacceptable toxicity or refusal to continue study treatment.
  Interventions: Drug: LAM561; Drug: TMZ; Radiation: RT

INTERVENTIONS:
Drug: LAM561 — Subjects in Arm B will receive orally LAM561 during the Chemoradiation Phase.
  Subjects in Arm B will receive LAM561 orally during the Maintenance (Adjuvant) Phase. Patients will continue to be administered with LAM561/Placebo after cycle 6 of the monotherapy phase until end of study. Adjuvant treatment will be discontinued upon determination of tumour progression as defined by RANO criteria, unacceptable toxicity, or refusal to continue study treatment.
  Arms: Arm B: SoC + 12 g/day of LAM561
Drug: TMZ — TMZ will be administered at 75 mg/m2, orally, once daily, continuously from Day 1 of radiotherapy to the last day of radiation for a maximum of 49 days.
  During the Maintenance (Adjuvant) Phase, all subjects will receive oral TMZ 150 - 200 mg/m2 once daily on Days 1 - 5 of each 28-day cycle for 6 cycles.
Radiation: RT — During the Chemoradiation Phase, all subjects will undergo focal RT, with one treatment given daily 5 days per week over approximately 6 weeks (and no more than 7 weeks).

SUMMARY:
The proposed Phase IIB/III randomized, double-blind, placebo-controlled trial in subjects with newly diagnosed primary glioblastoma multiforme (ndGBM) aims to compare the efficacy and safety of LAM561 versus placebo, given with standard of care (SoC) therapy of radiation therapy plus temozolomide (TMZ), followed by an adjuvant treatment of 6 month period of TMZ and then LAM561 or placebo in monotherapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 2 parallel arms (1:1 ratio), adjuvant trial to assess the efficacy of LAM561 versus placebo in patients with newly diagnosed, IDH1 wildtype, GBM. In all arms, patients will receive the SoC and will be randomized to receive either placebo or LAM561 dose.

The study is planned to enrol 140 patients. The primary endpoints of the study are PFS (for CMA) and OS (for FMA) as assessed after observing at least 66 PFS events and at least 90 OS events, respectively. It is expected that the analysis for PFS will be performed 1-2 years earlier than the analysis for OS.

An IDMC (Independent Data Monitoring Committee) meeting took place to assess the trial's futility and safety data from the start of the trial until September 2023. The IDMC had open access to the data without blinding; after analysis IDMC concluded that there were no concerns that would necessitate stopping the study for ethical reasons or safety issues that could adversely affect patients due to taking the medication, so the study is continuing as normal with no changes.

After 45 events for PFS are observed, a formal interim analysis will be performed and the data reviewed by an Independent Data Monitoring Committee (IDMC) or may be activated by the IDMC 12 months after the inclusion of the last patient if follow up is sufficient to identify an overall PFS or OS significant deviation from the literature. After reviewing the interim results, the iDMC will make recommendations regarding: the sample size and the continuation of the trial overall.

Further, the sample size and events will be re-estimated to ensure that the statistical power is maintained given the estimated treatment effect at interim analysis. The events/sample size increase will be based on the considerations of the success probability.

For that purpose, based on the conditional power, the interim results will be classified into the following zones: favourable, unfavourable or promising.

If the interim results fall in the promising zone, then it is planned to increase the total number of events both for PFS and OS by up to 50%, with up to 99 events for PFS and up to 135 events for OS. The total sample size will also be increased to up to 210 patients to ensure the desired number of events within a realistic time. If the interim results are favourable or unfavourable, the study size will remain as initially planned with 66 events for PFS and 90 for OS, collected from 140 patients.

The IDMC committee experts met in February 2024 after 45 PFS events occurred in the trial. Unblinded medical and clinical statistical data from 103 patients were evaluated to assess the efficacy - progression free survival (tumour growth or clinical deterioration) - of LAM561. The IDMC confirmed that, at the current level of evidence, after evaluating the Conditional Power of the unblinded results, no futility has been identified and recommends continuation of the study without modification.

In November 2024, After reaching 66 PFS events as stated by protocol, the independent data monitoring committee (IDMC) analyzed the data and recommended: (1) Continue the trial without modifications until 90 OS events (overall survival), when the final analysis will be carried out, estimated for Q4 2026; (2) that the trial should not be stopped for reasons of safety or futility and (3) opening the study, that is, removing the blind. From that moment, patients, doctors and Laminar as sponsor are able to know if any patient received placebo or LAM561.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent, signed and dated
2. Subjects who are able to understand and follow instructions during the trial
3. Age ≥18 and ≤75
4. Subjects with newly histologically confirmed intracranial malignant glioma (glioblastoma WHO Grade IV) that is IDH1 wildtype (local assessment) and who are scheduled to receive chemo-radiotherapy with temozolomide
5. Ability to swallow and retain oral medication
6. Centrally obtained MGMT promoter methylation status
7. Subjects who underwent total or partial / incomplete resection and with the appropriate quantity of tumour tissue releasable for eligibility
8. Karnofsky Performance Score (KPS) > 50 %
9. Female subjects with a childbearing potential must have a negative pregnancy test within one week before inclusion in the trial. Those female and male subjects admitted in the study must use a reliable method of contraception, for female subjects during the study period up until 32 days after last study treatment and for male subjects up until 92 days after last study administration.

   Women must be:
   * Either of NOT childbearing potential: postmenopausal (≥ 60 years of age, or < 60 years of age and amenorrhoea for 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression with follicle-stimulating hormone (FSH) above 40 U/L and oestradiol below 30 ng/L, or if taking tamoxifen or toremifene, and age < 60 years, then FSH and oestradiol in the postmenopausal range), permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy), or otherwise incapable of pregnancy
   * Or of childbearing potential and practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; male partner sterilization (the vasectomized partner should be the sole partner for that subject).
10. A man who is sexually active and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom or partner with occlusive cap (diaphragm or cervical/vault caps).
11. Adequate bone marrow function including: Absolute neutrophil count (ANC) ≥1,500/mm^3 or ≥1.5 x 10^9/L; Platelets ≥ 100,000/mm3 or ≥100 x10^9/L; Haemoglobin ≥ 9 g/dL (may have been transfused).
12. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal range (ULN), an aspartate aminotransferase (AST), level ≤ 2.5 × ULN, and an alanine aminotransferase (ALT) level ≤ 2.5 × ULN or, for subjects with documented metastatic disease to the liver, AST and ALT levels ≤ 5 × ULN. Subjects with documented Gilbert disease are allowed if total bilirubin ≤ 3 x ULN
13. Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula

Exclusion Criteria:

1. Known hypersensitivity to any component of the investigational product.
2. Any other investigational drug within the preceding 30 days. Prior, concomitant, or planned concomitant treatment with anti-neoplastic aim including (but not limited) to NovoTumor Treatment Fields (Novo TTF), bevacizumab, intratumoural or intracavitary anti-neoplastic therapy (e.g Gliadel wafers), or other experimental therapeutics intended to treat the tumour.
3. Subjects who underwent "only biopsy" resection
4. Anticancer therapy within 4 weeks of study entry (6 weeks for mitomycin and nitrosoureas)
5. Other major surgery within the preceding 30 days
6. Allergy, hypersensitivity or other intolerability to temozolomide and its excipients, patients with hypersensitivity to dacarbazine and patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
7. Unable to undergo MRI
8. Presenting with diffuse midline gliomas or multifocal GBM (distant from the flare or contralateral) or rapid progression between early post-surgery MRI and pre-radiotherapy MRI
9. Uncontrolled or significant cardiovascular disease
10. A history of uncontrolled hyperlipidaemia and/or the need for concurrent lipid lowering therapy
11. Need for warfarin, phenytoin or sulphonylureas (glibenclamide, glimepiride, glipizide, glyburide or nateglanide)
12. Past medical history of uncontrolled clinically significant active or chronic gastrointestinal disorders (for example, Crohn's disease, celiac disease, untreated stomach ulcers, etc) and gastro-inflammatory pathologies
13. Uncontrolled diabetes mellitus, with glycated haemoglobin (HbA1c) levels at the screening visit of ≥7.5%
14. Cardiac disease, defined specifically as either

    1. Mean resting corrected QT interval (QTc) > 470 msec (for women) and > 450 ms (for men) obtained from 3 consecutive ECGs
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (example, complete left bundle branch block, third degree heart block)
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, potential for Torsades de Pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age
15. Previous malignancies within the last three years other than ndGBM, except successfully treated squamous cell carcinoma of the skin, superficial bladder cancer, and in situ carcinoma of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of LAM561 in combination with the standard of care (SoC) treatment of radiotherapy (RT) and TMZ. | Assessed after observing at least 66 PFS events
  To evaluate the efficacy of LAM561 in combination with the standard of care (SoC) treatment of radiotherapy (RT) and TMZ, as assessed by
  - Progression Free Survival (PFS) using the Response Assessment in Neuro-Oncology (RANO) criteria
To evaluate the efficacy of LAM561 in combination with the standard of care (SoC) treatment of radiotherapy (RT) and TMZ. | Assessed after observing at least 90 OS events
  To evaluate the efficacy of LAM561 in combination with the standard of care (SoC) treatment of radiotherapy (RT) and TMZ, as assessed by
  - Overall Survival (OS)

SECONDARY OUTCOMES:
To evaluate measures of clinical response | Baseline and Post-baseline: day 1 of each odd cycle of maintenance/monotherapy phase and at progression
  Changes in neurological function, based on Neurologic Assessment in Neuro-Oncology (NANO) criteria
To evaluate additional measures of efficacy | Baseline and Post-baseline: day 1 of each odd cycle of maintenance/monotherapy phase and at progression
  Time to Progression (TTP) (as assessed using RANO criteria)
To characterize the pharmacokinetics (PK) and pharmacodynamics (PD) parameters | At week 3 and 5 (day in both cases) of chemo-radiotherapy phase and at day 1 and 15 of cycle 1 of the maintenance phase
  Blood samples for determination of plasma concentrations of LAM561 in combination with RT and/or TMZ.
  Maximum Plasma Concentration [Cmax]
To characterize the pharmacokinetics (PK) and pharmacodynamics (PD) parameters | At week 3 and 5 (day in both cases) of chemo-radiotherapy phase and at day 1 and 15 of cycle 1 of the maintenance phase
  Blood samples for determination of plasma concentrations of LAM561 in combination with RT and/or TMZ.
  Lowest plasma concentration reached before the next dose is administered (Trough)
To characterize the pharmacokinetics (PK) and pharmacodynamics (PD) parameters | At week 3 and 5 (day in both cases) of chemo-radiotherapy phase and at day 1 and 15 of cycle 1 of the maintenance phase
  Blood samples for determination of plasma concentrations of LAM561 in combination with RT and/or TMZ.
  Area Under the plasma concentration-time Curve (AUC)
To evaluate Health-related Quality of Life (HRQoL) | Baseline and Post-baseline: day 1 of each odd cycle of maintenance/monotherapy phase and at progression
  HRQoL assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, EORTC-QLQ C30, version 3.0 and brain cancer specific QLQ-BN20.
  The QLQ-C30 is a 30-item patient self-report questionnaire composed of both multi-item and single scales, including five functional scales (physical, role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status/HRQoL scale, and six single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties). Subjects rate items on a four-point scale, with 1 as "not at all" and 4 as "very much". The QLQ-C30 was developed and validated for use in a cancer patient population, and its reliability and validity is highly consistent across different language-cultural groups.
To evaluate Health-related Quality of Life (HRQoL) | Baseline and Post-baseline: day 1 of each odd cycle of maintenance/monotherapy phase and at progression
  HRQoL assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, EORTC-QLQ C30, version 3.0 and brain cancer specific QLQ-BN20.
  The QLQ-BN20 is a 20-item patient self-report questionnaire that was developed specifically as a module for subjects with brain cancer. It consists of four domain scores, including future uncertainty, visual disorder, motor dysfunction, and communication deficit, as well as seven individual symptom items (headache, seizures, drowsiness, hair loss, itching, difficulty with bladder control, and weakness of both legs). Subjects rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A retrospective validation study has been conducted confirming its psychometric validity.
To evaluate Health-related Quality of Life (HRQoL) | Baseline and Post-baseline: day 1 of each odd cycle of maintenance/monotherapy phase and at progression
  HRQoL assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, EORTC-QLQ C30, version 3.0 and brain cancer specific QLQ-BN20.
  The EORTC QLQ-C30/BN20 as outlined in SoA. These assessments should be completed prior to study drug administration and any other study procedures being performed at these visits, and prior to discussing with the subject that their disease has progressed.

CONTACTS AND LOCATIONS:
Locations (22):
- France (4):
  - Institut Cancerologie de L'Ouest (ICO), Angers
  - Centre Eugène Marquis (CEM), Rennes
  - Gustave Roussy University Hospital, Rennes
  - Institut universitaire du cancer, Toulouse
- Reaserch Fund of the Hadassah Medical Organization, Jerusalem, Israel
- Italy (4):
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - Istituto Nazionale Tumori "Regina Elena", Roma
  - University of Turin, Turin
- Spain (9):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitari i Politécnic La Fe., Valencia, Valencia
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Parc Tauli, Sabadell
- United Kingdom (4):
  - Freeman Hospital's Northern Centre of Cancer Care, Newcastle, Newcastle Upon Tyne
  - University Hospitals Birmingham NHS Foundation Trust - New Queen Elizabeth Hospital, Birmingham
  - Cambridge university hospital, Cambridge
  - The Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided